CLINICAL TRIAL: NCT03653962
Title: Video-Assisted Presentation Before Bariatric Surgery Enhanced Understanding of Informed Consent Content: Randomized Controlled Trial
Brief Title: Video-Assisted Presentation Before Bariatric Surgery Enhanced Understanding of Informed Consent Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Kutay Saglam, MD, Gastrointestinal Surgery Fellow, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kutay Saglam
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Bariatric Surgery Candidate
Keywords: Multimedia; informed consent; metabolic surgery; Roux-en-Y gastric bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- only informed consent (Active Comparator): The first group was given verbal-written informed consent and a 15 question quiz about the informed consent content afterwards.
  Interventions: Behavioral: non-video group
- video assisted group (Experimental): The second group got an additional information video presentation and then the same quiz.
  Interventions: Behavioral: video assisted group; Behavioral: non-video group

INTERVENTIONS:
Behavioral: video assisted group
  Arms: video assisted group
Behavioral: non-video group

SUMMARY:
This study evaluates the addition of video presentation on conventional informed consent. Participants divided two randomly, one group read only conventional informed consent, the other video presentation was watched after reading conventional consent.

ELIGIBILITY:
Inclusion Criteria:

* being a being bariatric metabolic surgery candidate according to international guidelines

Exclusion Criteria:

* illiterate
* previous bariatric surgery
* age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Questionnaire | six months
  In the video group : verbal-written consent + video presentation In the conventional consent group: only verbal-written consent
  The video consisted of a summary of the written informed consent. Questionnaire consist of 15 questions quiz was given to both groups. Each question was rated on 15 points. 1point = bad score means don't understand informed consent. 15 point = full score means good understanding.

IPD SHARING:
Plan to Share IPD: No